CLINICAL TRIAL: NCT06868979
Title: Optical Imaging as a Diagnostic Tool for Monitoring Brain Function in X-linked Rare Disorders
Brief Title: Optical Imaging in X-linked Disorders.
Acronym: IMAGINER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL23_0409; 2024-A01730-47 (Other: ID-RCB)
Record Dates: First submitted 2025-02-14; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Fragile X Syndrome (FXS); Creatine Transporter Deficiency
Keywords: Fragile X syndrome; Optical imaging; brain function; Creatine transporter; cognitive function; reasoning tasks
MeSH Terms: conditions — Fragile X Syndrome; Creatine deficiency, X-linked | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Intervention Model Description: This is a multicentric prospective, cross-sectional case control study to determine biomarkers to be used in future clinical trials in CTD and FXS patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CTD (Creatine Transporter Deficiency ) patients (Other): Male CTD patients having a confirmed mutation in the SLC6A8 gene, aged > 5 to < 35 years.
  Interventions: Other: Clinical assessment; Other: Parental questionnaires; Other: Cognitive assessment; Other: Reasoning assessment; Device: fNIRS assessement
- FXS (Fragile X Syndrome) patients (Other): Male FXS patients having a confirmed full mutation in the FMR1 gene (>200 GCC repeats), aged > 5 to < 35 years.
  Interventions: Other: Clinical assessment; Other: Reasoning assessment; Device: fNIRS assessement
- Chronological age-matched controls (Other): Male aged > 5 to < 35 years.
  Interventions: Other: Clinical assessment; Other: Parental questionnaires; Other: Cognitive assessment; Other: Reasoning assessment; Device: fNIRS assessement

INTERVENTIONS:
Other: Clinical assessment — Clinical examination including Medical history, developmental trajectory, epilepsy history, ASD symptoms, clinical examination at the inclusion visit by a neuropediatrist
Other: Parental questionnaires — Parental questionnaires including Vineland-2, ABC, CBCL, PPD-MRS, SRS-2 and BRIEF completed at the inclusion visit
  Arms: CTD (Creatine Transporter Deficiency ) patients; Chronological age-matched controls
Other: Cognitive assessment — Cognitive assessment including Leiter-3, PPVT 5, EVT 3 completed at the inclusion visit
  Arms: CTD (Creatine Transporter Deficiency ) patients; Chronological age-matched controls
Other: Reasoning assessment — Simple reasoning tasks on tablets performed at the inclusion visit.
Device: fNIRS assessement — Imaging session using fNIRS (NIRSport 8x8, NIRx Medical Technologies LLC, Berlin, Germany) performed at the inclusion visit.

SUMMARY:
Fragile X syndrome (FXS, OMIM #300624) and Creatine Transporter Deficiency (CTD, #300352) are the two most common causes of X-linked intellectual disability. FXS and CTD affect hemizygous males and with highly variable severity heterozygous females. Both these neurodevelopmental disorders (NDDs) have a dramatic impact on the family quality of life and the health-care system. These disorders share common clinical traits, including intellectual disability, autistic-like features, behavioural and mood alterations and seizures. Brain anatomy appears largely normal, suggesting that functional deficits result from subtle changes in synaptic connectivity. Moreover, common physiological mechanisms related to brain energetics might concur to the pathophysiology of FXS and CTD. Indeed, FMR1 and SLC6A8 are directly involved in the regulation of metabolism and the loss-of-function of both genes leads to a disruption of the mitochondrial network.

There is no cure for these disorders and the efficacy study of potential treatments is hindered by the scarcity of unbiased, quantitative, non-invasive biomarkers for monitoring brain function.

This is a critical problem, since the often-used phenotypic observation of behavioural endpoints to score NDDs such as FXS and CTD is highly prone to subjective bias. For successful clinical trials, the availability of objective readouts is crucial to evaluate the therapeutic response to new drugs. There are multiple techniques to visualize neural circuit activity in the living brain. Interestingly, FXS and CTD are the only two NDDs that at preclinical level show an abnormally large hemodynamic response to sensory stimulation in functional imaging studies of intrinsic optical signals.

The objective of this project is to exploit optical imaging techniques to devise a measurable and non-invasive biomarker of brain function in FXS and CTD. Since a disruption of brain energy metabolism is a major disease mechanism linking these disorders, we hypothesized that the assessment of the cerebral blood flow and oxygen consumption represents a sensitive readout for quantifying functional alterations of neural circuits.

Functional near-infrared spectroscopy (fNIRS), allows quantifying changes of hemoglobin species and local blood flow in the cerebral cortex of humans, providing an indirect measure of neuronal activity. In the clinical framework, this blood-oxygen-level-dependent signal is similar to that detected with functional MRI (fMRI). However, fNIRS has the advantage of being completely non-invasive, low-cost, portable, noiseless, endowed with high experimental flexibility and easy to implement in both laboratory and clinical settings. Moreover, fNIRS is more tolerant to motion artifacts than fMRI, and robust methods for motion detection/correction allow to image very young children without sedation. These methodological strengths make fNIRS as an outstanding choice for investigating neural circuits in clinically relevant populations at the very-low cost. Although introduced into the clinical care almost 40 years ago, fNIRS gained much popularity in the study of brain development and NDDs only recently. To date, however, fNIRS has been used primarily to investigate the typical maturation of speech perception and language, sensory and motor functions, social communication and interaction, object and action processing in toddlers and children.

In this proposal, the investigators hypothesize that by combining the above-mentioned strengths of fNIRS to the clinical study of several cognitive and motor parameters, the investigators can define unique "fNIRS signatures" for FXS and CTD as brain biomarkers for the diagnosis and the assessment of treatment outcomes. Since the measurement of visual responses has been introduced as a quantitative method to assess brain function in NDDs, the investigators will test the value of visually-evoked fNIRS signals in classifying patients and predicting symptom severity in the FXS and CTD clinical population. Preliminary data in the mouse models of CTD and FXS strongly suggest that visual hemodynamic responses (vHDR) are markedly altered in the occipital cortex of mutant animals. Morever, the investigators will use a standardized procedure with high entertaining value to measure vHDR in the occipital cortex of children.

ELIGIBILITY:
Inclusion Criteria :

CTD patients :

* male
* having a confirmed mutation in the SLC6A8 gene
* ≥ 5 to ≤ 35 years old
* whose maternal language is French,
* having signed the informed consent and/or for whom parents (for children)/legal guardian (for protected adults) have signed the informed consent.
* affiliated to national Health Insurance system (sécurité sociale) or parents/legal guardian affiliated to national health insurance system

FXS patients :

* male
* having a confirmed full mutation in the FMR1 gene (>200 GCC repeats)
* ≥ 5 to ≤ 35 years old
* whose maternal language is French,
* having signed the informed consent and/or for whom parents (for children)/legal guardian (for protected adults) have signed the informed consent.
* affiliated to national Health Insurance system (sécurité sociale) or parents/legal guardian affiliated to national health insurance system

Chronological age-matched controls :

* male
* ≥ 5 to ≤ 35 years old
* whose maternal language is French,
* having signed the informed consent and/or for whom parents have signed the informed consent.
* affiliated to national Health Insurance system (sécurité sociale) or parents/legal guardian affiliated to national health insurance system

Exclusion Criteria:

CTD patients :

* Refusal of the subject and/or the subject's parents/legal guardian to sign the informed consent
* Refusal of the subject and/or the subject's parents/legal guardian to be informed of possible abnormalities detected during the neuropsychological assessment.

FXS patients :

* Refusal of the subject and/or the subject's parents/legal guardian to sign the informed consent
* Refusal of the subject and/or the subject's parents/legal guardian to be informed of possible abnormalities detected during the neuropsychological assessment.

Chronological age-matched controls :

* Refusal of the subject and/or the subject's parents/legal guardian to sign the informed consent
* Refusal of the subject and/or the subject's parents/legal guardian to be informed of possible abnormalities detected during the neuropsychological assessment.
* History of neurological or psychiatric disorder,
* Repetition of a grade,
* Learning disability requiring rehabilitation (speech therapy, psychomotor or oculomotor therapy).

Ages: 5 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Amplitude of the visual hemodynamic response | Inclusion visit
  Cortical hemodynamic activity data recorded via fNIRS imaging in response to visual stimulation (task-evoked) using a cartoon-based stimulus. Measure of the amplitude of the peak response to viewing radial checkerboard blended with the animated cartoon for total Hb, OxyHb and DeoxyHb concentration change.
Latency of the visual hemodynamic response | Inclusion visit
  Cortical hemodynamic activity data recorded via fNIRS imaging in response to visual stimulation (task-evoked) using a cartoon-based stimulus. Measure of the latency of the peak response to viewing radial checkerboard blended with the animated cartoon for total Hb, OxyHb and DeoxyHb concentration change.

SECONDARY OUTCOMES:
Clinical Endpoints_Presence of epilepsy | Inclusion visit
  Presence of epilepsy
Clinical Endpoints_Type of epilepsy | Inclusion visit
  Type of epilepsy
Clinical Endpoints_Treatment of epilepsy | Inclusion visit
  Antiepileptic treatment (if any)
Clinical endpoints_Developmental trajectory | Inclusion visit
  Age at walking, Age at first words, Age at 2 words association, Age at first sentences
Clinical endpoints_Autism spectrum disorder (ASD) | Inclusion visit
  Autism spectrum disorder (ASD) diagnosis (using DSM5 criteria)
Cognitive assessment with Leiter 3 scale | Inclusion visit
  Score of the cognitive assessment obtained with the Leiter 3 scale (4 cognitive sub-tests to be able to compute the non-verbal IQ and 2 non-verbal memory sub-tests)
Cognitive assessment with Bayley 4 scale | Inclusion visit
  Score of the cognitive assessment obtained with Bayley 4 scale (if Leiter 3 scale is not possible)
Language assessment with the PPVT-5 test | Inclusion visit
  Score obtained with the PPVT-5 (Peabody Picture Vocabulary Test Fifth Edition) test for receptive vocabulary
Language assessment with the EVT-3 test | Inclusion visit
  Score obtained with the EVT-3 (Expressive Vocabulary Test third edition) test for expressive vocabulary.
Reasoning tasks | Inclusion visit
  Simple reasoning tasks on tablet (with four difficulty levels, A to D: match-to-sample task, categorization task, analogical reasoning task, implicit rules tasks). Reaction Time (RT) and Error Rate (ER) will be anayzed for each of the four reasoning tasks. The RT is defined as the time elapsing between the display of the image and the time when the subject selected one of the two answers.
Parental questionnaires to assess adaptive abilities (Vineland 2) | Inclusion visit
  Parental questionnaires to assess adaptive abilities (Vineland 2)
Parental questionnaires to assess behavioral disorder (ABC 2) | Inclusion visit
  Parental questionnaires to assess behavioral disorder (ABC 2)
Parental questionnaires to assess behavioral disorder (CBCL) | Inclusion visit
  Parental questionnaires to assess behavioral disorder (CBCL)
Parental questionnaires to assess autistic features (PDD-MRS) | Inclusion visit
  Parental questionnaires to assess autistic features (PDD-MRS)
Parental questionnaires to assess autistic features (SRS2) | Inclusion visit
  Parental questionnaires to assess autistic features (SRS2)
Parental questionnaires to assess executive functions (BRIEF) | Inclusion visit
  Parental questionnaires to assess executive functions (BRIEF)

CONTACTS AND LOCATIONS:
Locations (1):
- Woman, mother and child hospital, Hospices Civils de Lyon, Bron, France